CLINICAL TRIAL: NCT01612689
Title: 3-Dimensional Accelerometer Sub-Study for Patients Participating in the E-30 Study: Heart Rate Changes in Subjects With Epilepsy During an Epilepsy Monitoring Unit Admission
Brief Title: 3-Dimensional Accelerometer Sub-Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: E-30-S
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Epilepsy
Keywords: Accelerometer; EMU; Ambulatory; ECG; Heart rate
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physiologic Data Collection (Experimental)
  Interventions: Device: Accelerometer Device

INTERVENTIONS:
Device: Accelerometer Device — A sensor platform that enables physiological monitoring in routine, home or office environments.

SUMMARY:
This is a prospective, unblinded sub-study to the E-30 to gather physiological data.

DETAILED DESCRIPTION:
This sub-study to the E-30 is designed to collect vital signs, accelerometer and ECG data on subjects, and will consist of two phases. Phase 1 is designed to collect data in an Epilepsy Monitoring Unit (EMU) and Phase 2 is designed to collect data in an everyday (ambulatory) setting.

ELIGIBILITY:
Inclusion Criteria:

(Phase 1)

* Subject be scheduled to participated in the E-30 parent study for a minimum of 48 hours
* Subject has a clinical diagnosis of epilepsy based on a prior EMU visit

(Phase 1&2)

* Subject is currently enrolled or previously participated in the E-30 study
* Subject must be 6 years of age or older

(Sleep State: Optional)

* Subject must be 12 years of age
* Subject is currently enrolled in the E-30S sub-study and is willing to stay in a light controlled environment in the EMU for up to 120 hours

Exclusion Criteria:

(Phase 1&2)

* Subjects with a medical condition that in the opinion of the investigator would affect his/her ability to participate in the sub-study.
* Subject who has implanted defibrillator, pacemaker or Vagus Nerve Stimulation Therapy® (VNS) System
* Subjects who are pregnant or lactating
* Subjects with severe psychiatric disease that in the opinion of the investigator would prevent the subject's successful completion of the sub-study.
* Subjects 6 to 16 years of age with moderate/severe learning difficulties or those who may be at risk of self-harm.
* Subjects prescribed drugs specifically for a cardiac or autonomic disorder that in the investigator's opinion would affect heart rate response unless the patient has ictal tachycardia while taking said drugs. These include, but are not limited to, beta adrenergic antagonists ("beta blockers").
* Subjects with cardiovascular arrhythmias or cardiac disease that would preclude the ability to detect intrinsic changes in heart rate due to activity, stress, or seizure. This would include but not be limited to chronic atrial fibrillation or chronotropic incompetence.
* Subjects with a history of dependence on alcohol or narcotic drugs within the past 2 years as defined by DSM IV-R.

(Sleep State: Optional)

* Subjects with a history if gastrointestinal disease (GI)or GI surgery
* Subjects with a history of difficulty swallowing
* Subjects with diabetes mellitus
* Subjects with uncontrolled hypertension
* Subjects with planned MRI during EMU stay

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Gather physiological data | Up to 2 weeks
  The purpose of this sub-study is to gather physiological data in consenting subjects who were previously enrolled in the "parent" E-30 study (NCT01202669).

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Olin, Study Director — Cyberonics, Inc.
Locations (2):
- United States (2):
  - Gainesville, Florida
  - Chicago, Illinois